CLINICAL TRIAL: NCT03932929
Title: 36-Month Clinical Evaluation of Different Adhesive Strategies of a Universal Adhesive
Brief Title: 36-Month Clinical Evaluation of a Universal Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Cansu Atalay, Pricipal Investigator, DDS, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KA-17088
Record Dates: First submitted 2019-04-17; First posted 2019-05-01 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Non-Carious Cervical Lesions
Keywords: Non-Carious Cervical Lesions; Universal adhesive

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scotchbond universal adhesive (etch-and-rinse) (Experimental): Acid etch (enamel&dentin)+adhesive agent Intervention: Device: Adhesive agent
  Interventions: Device: Scotchbond Universal Adhesive (3M ESPE)
- Scotchbond universal adhesive (selective-etch) (Experimental): Acid etch (only enamel)+adhesive agent Intervention: Device: Adhesive agent
  Interventions: Device: Scotchbond Universal Adhesive (3M ESPE)
- Scotchbond universal adhesive (self-etch) (Experimental): Adhesive agent Intervention: Device: Adhesive agent
  Interventions: Device: Scotchbond Universal Adhesive (3M ESPE)

INTERVENTIONS:
Device: Scotchbond Universal Adhesive (3M ESPE) — Adhesive system

SUMMARY:
The aim of this clinical trial was to evaluate and compare the performance of a universal adhesive with different adhesive strategies in the restoration of non-carious cervical lesions (NCCLs) over a 36-month period.

DETAILED DESCRIPTION:
One hundred sixty-five NCCLs in 35 patients (13 female, 22 male) with at least 3 lesions were included in this study. Three groups were formed according to adhesive strategies used (n=55): selective-etch mode; etch-and-rinse mode (ER); or self-etch (SE) mode of a universal adhesive, Single Bond Universal. The same nanofilled resin composite, Filtek Ultimate was used for all restorations by a single operator. The restorations were evaluated by two calibrated examiners at baseline and at 6-, 12-, 18-, 24- and 36- months in accordance with the modified USPHS criteria. The Chi-square test was used for intergroup, the Cochran Q test was used for intragroup comparison.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* good oral hygiene
* available for recall
* at least 20 teeth under occlusion
* the presence of at least three non-carious cervical lesions

Exclusion Criteria:

* poor oral hygiene
* bruxism habits
* severe or chronic periodontitis
* If the teeth selected for study, were nonvital, or had any restorations on other surfaces were not included.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-09-02 (Actual)

PRIMARY OUTCOMES:
Marginal adaptation | From baseline to 36 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal adaptation. Marginal adaptation was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed . Scores; Alfa: Closely adapted, no visible crevice. Bravo: Visible crevice, explorer will penetrate. Charlie: Crevice in which dentin is exposed
Marginal staining | From baseline to 36 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal staining. Marginal staining was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed . Scores: Alfa: No discoloration. Bravo: Discoloration without. Charlie: Discoloration with penetration in pulpal direction
Retention | From baseline to 36 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by 2 independent clinicians. Scores: Alfa: No loss of restorative material. Charlie: Any loss of restorative material
Postoperative sensitivity | From baseline to 36 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by 2 independent clinicians. Scores: Alfa: Not present. Bravo: sensitive but diminishing in intensity. Charlie:constant sensitivity, not diminishing in intensity
Seconder caries | From baseline to 36 month
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by 2 independent clinicians. Scores: Alfa: No caries present. Charlie: Caries present

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lawson NC, Robles A, Fu CC, Lin CP, Sawlani K, Burgess JO. Two-year clinical trial of a universal adhesive in total-etch and self-etch mode in non-carious cervical lesions. J Dent. 2015 Oct;43(10):1229-34. doi: 10.1016/j.jdent.2015.07.009. Epub 2015 Jul 29. PMID 26231300
- [Background] Hanabusa M, Mine A, Kuboki T, Momoi Y, Van Ende A, Van Meerbeek B, De Munck J. Bonding effectiveness of a new 'multi-mode' adhesive to enamel and dentine. J Dent. 2012 Jun;40(6):475-84. doi: 10.1016/j.jdent.2012.02.012. Epub 2012 Feb 28. PMID 22381614
- [Background] Perdigao J, Kose C, Mena-Serrano AP, De Paula EA, Tay LY, Reis A, Loguercio AD. A new universal simplified adhesive: 18-month clinical evaluation. Oper Dent. 2014 Mar-Apr;39(2):113-27. doi: 10.2341/13-045-C. Epub 2013 Jun 26. PMID 23802645